CLINICAL TRIAL: NCT06430450
Title: Determination of Salivary Soluble Urokinase Plasminogen Activator Receptor (SuPAR), Hypoxia-inducible Factor-1 Alpha (HIF-1α), E-cadherin, Galectin 3, IL-4, IL-10 and TNF-α Levels in Individuals With Different Degrees of Periodontal Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, İsmail Taşdemir, Assistant professor, Karamanoğlu Mehmetbey University
Other Study IDs: ISMAILKMU
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: Periodontitis; Saliva; Cytokine
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healty: Individuals who have no clinical signs of inflammation in the periodontal tissues and the number of areas showing bleeding on probing does not exceed 20%.
  Interventions: Diagnostic Test: Clinical measurements and saliva samples collection
- Grade A: Individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant of the jaw, attachment loss, and radiological bone loss percentage/age ratio in the tooth with the most bone loss <0.25
  Interventions: Diagnostic Test: Clinical measurements and saliva samples collection
- Grade B: Individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant jaw, attachment loss, and a radiological bone loss percentage/age ratio of 0.25-1.0 in the tooth with the most bone loss.
  Interventions: Diagnostic Test: Clinical measurements and saliva samples collection
- Grade C: Individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant of the jaw, attachment loss, and a radiological bone loss percentage/age ratio >1.0 in the tooth with the most bone loss.
  Interventions: Diagnostic Test: Clinical measurements and saliva samples collection

INTERVENTIONS:
Diagnostic Test: Clinical measurements and saliva samples collection — Clinical measurements will be taken from all patients and saliva samples will be collected for biochemical analysis.

SUMMARY:
The aim of this clinical study is; Comparatively comparing salivary Soluble Urokinase Plasminogen Activator Receptor (SuPAR), Hypoxia-inducible factor-1 alpha (HIF-1α), E-cadherin, galectin 3, IL-4, IL-10 and TNF-α levels in individuals with different Periodontal Disease Degrees and to evaluate and analyze correlations with clinical parameters. In our study, saliva samples will be taken from a total of 80 systemically healthy volunteers, 20 of patients are periodontal healthy, 20 of patients have degree A periodontitis, 20 of patients have degree B periodontitis and 20 of patients have degree C periodontitis, along with the measurement of whole mouth clinical parameters. Soluble Urokinase Plasminogen Activator Receptor (SuPAR), Hypoxia-inducible factor-1 alpha (HIF-1α), E-cadherin, galectin 3, IL-4, IL-10 and TNF-α levels in the samples taken will be subjected to enzyme-related immunoassay ( It will be determined by ELISA). Cytokine levels between different groups will then be interpreted as a result of statistical analysis. Possible significant differences shed light on future studies with Soluble Urokinase Plasminogen Activator Receptor (SuPAR), Hypoxia-inducible factor-1 alpha (HIF-1α), E-cadherin, galectin 3, IL-4, IL-10 and TNF-α. These cytokines may help develop different diagnostic methods or treatment strategies in future periodontal treatments.

DETAILED DESCRIPTION:
The study included patients between the ages of 18 and 70 who applied to Karamanoğlu Mehmetbey University Ahmet Keleşoğlu Faculty of Dentistry Department of Periodontology, were non-smokers, had no systemic problems, had not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 3 months, were not pregnant, had not received periodontal treatment in the last 6 months, and having at least 20 teeth in its mouth; for grade A periodontitis group; 20 individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant of the jaw, attachment loss, and radiological bone loss percentage/age ratio <0.25 in the tooth with the most bone loss; for grade B periodontitis group; 20 individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant jaw, attachment loss, and a radiological bone loss percentage/age ratio of 0.25-1.0 in the tooth with the most bone loss; for grade C periodontitis group; 20 individuals with a probing pocket depth of 5 mm or more in at least 2 teeth in each quadrant of the jaw, attachment loss, and radiological bone loss percentage/age ratio >1.0 in the tooth with the most bone loss; For the healthy group; According to the evaluation made in 6 regions of each tooth, including 20 individuals who show bleeding on probing in less than 20% of the area, have a probing depth of less than 4 mm, and have no attachment loss. The healthy and periodontal disease group will consist of 80 patients in total.Anamnesis will be taken from individuals at the beginning of the interview, and individuals who meet the specified criteria after the anamnesis will be included in the study. After being informed about the study, an informed consent form will be obtained from the individuals.

After the anamnesis is taken, clinical periodontal evaluations will be performed on individuals who are deemed to meet the inclusion criteria. Clinically, plaque index (Sillness and Löe 1964), gingival index (Löe and Sillness 1963), pocket depth and bleeding on probing index(Ainamo&Bay, 1975) will be recorded.

Saliva samples will be taken from individuals divided into groups for biochemical examinations. Saliva samples will be taken from each patient, first frozen at -20ºC and than stored at -28ºC until the day of analysis. Cytokine levels in the samples collected from the patients will be determined by the enzyme-related immune test "Enzyme Linked-Immuno-Sorbent Assay" (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a varying degree of periodontal status (periodontally healthy, gingivitis, and chronic periodontitis).
* Have no systemic disease.
* No smoking/ not using any tobacco products or alcohol.
* No periodontal therapy in last 6 months.
* Not using any anti-inflammatory drugs in last 3 months and antibiotics in last 6 months.
* Not to be pregnant or in lactation period.
* Having ≥20 permanent teeth.

Exclusion Criteria:

* Having any systemic disease.
* Smokers, other tobacco product, and alcohol consumers.
* Having any periodontal therapy in last 6 months.
* Using any anti-inflammatory drugs in last 3 months and antibiotics in last 6 months.
* Being pregnant or in lactation period.
* Having ˂20 permanent teeth.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 20 healty patients
  * 20 Grade A periodontitis
  * 20 Grade B periodontitis
  * 20 Grade C periodontitis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | First 5 months
  Comparatively comparing salivary Soluble Urokinase Plasminogen Activator Receptor (SuPAR), Hypoxia-inducible factor-1 alpha (HIF-1α), E-cadherin, galectin 3, IL-4, IL-10 and TNF-α levels in individuals with different Periodontal Disease Degrees. To examine and determine the correlation of these cytokines with clinical measurements.

SECONDARY OUTCOMES:
Outcome 2 | Two months after the study was completed
  By investigating the changes in these cytokine levels in the presence of periodontal disease, they can be used in disease diagnosis in the future or to provide preliminary information on possible treatments that can be performed through these cytokine pathways.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tasdemir I, Ozgoren O, Yilmaz HE, Kartal E, Altunyaprak S, Saglam M. Salivary levels of suPAR, HIF-1alpha and TNF-alpha in different grades of stage III periodontitis. BMC Oral Health. 2025 May 22;25(1):760. doi: 10.1186/s12903-025-06155-3. PMID 40405145